CLINICAL TRIAL: NCT01443793
Title: Longitudinal Pattern of Streptococcus Pneumoniae Nasopharyngeal Carriage and Antimicrobial Susceptibility in Healthy Children Aged Less Then 5 Years, in the Area of Milan and Surroundings, Lombardy, Italy.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Gian Vincenzo Zuccotti, professor of Pediatrics, University of Milan
Other Study IDs: Pneumo01
Record Dates: First submitted 2011-09-28; First posted 2011-09-30 (Estimated); Last update posted 2011-10-04 (Estimated); Status verified 2011-10

CONDITIONS: Streptococcus Pneumoniae Nasopharyngeal Carriage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this active surveillance study is to make available crucial data about epidemiology, serotype distribution, and longitudinal pattern of antibiotic susceptibility of nasopharyngeal strains of Streptococcus pneumoniae carried in the population of healthy children aged less than years and living in the area of Milan and surroundings, Lombardy, Italy.

* To estimate the nasopharyngeal carriage rate and longitudinal pattern of Streptococcus pneumoniae in healthy children aged less than 5 years living in the area of Milan, Italy;
* To describe the circulation of antimicrobial non-susceptible Streptococcus pneumoniae strains in healthy children aged less than 5 years

Secondary objectives:

* To describe the nasopharyngeal carriage distribution of Streptococcus pneumoniae strains in healthy subjects less than 5 years old;
* To examine the role of risk factors in the Streptococcus pneumoniae carriage rate in healthy children;
* • To evaluate the possible impact of vaccination policy in the referenced population.

ELIGIBILITY:
Inclusion Criteria:

* To estimate the nasopharyngeal carriage rate and longitudinal pattern of Streptococcus pneumoniae in healthy children aged less than 5 years living in the area of Milan, Italy;
* To describe the circulation of antimicrobial non-susceptible Streptococcus pneumoniae strains in healthy children aged less than5 years

Exclusion Criteria:

* To describe the nasopharyngeal carriage distribution of Streptococcus pneumoniae strains in healthy subjects less than 5 years old;
* To examine the role of risk factors in the Streptococcus pneumoniae carriage rate in healthy children;
* To evaluate the possible impact of vaccination policy in the referenced population..

Ages: 3 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The sample size is calculated to detect at baseline at least 100 nasopharyngeal swab specimens positive for Streptococcus pneumoniae, and possibly further 100 positive swabs at both 6 and 12 months after recruitment. A probability sample of at least 1,300 children will be recruited. Children will be selected using a randomization list of assisted children less than 5 years-old that will be computer generated for any of participant Family Pediatrician, based on the Lombardy Regional Health Databases and using the National Insurance Number.
Sampling Method: Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2011-09

PRIMARY OUTCOMES:
• circulation of antimicrobial non-susceptible Streptococcus pneumoniae strains in healthy children aged less than 5 years | 1 year

SECONDARY OUTCOMES:
• the nasopharyngeal carriage distribution of Streptococcus pneumoniae strains in healthy subjects less than 5 years old; | 1 year
• the role of risk factors in the Streptococcus pneumoniae carriage rate in healthy children; | 1 year
• the possible impact of vaccination policy in the referenced population | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- AO L.Sacco, Milan, Italy, Italy